CLINICAL TRIAL: NCT04282980
Title: A Multicenter Phase 2, Single-Arm Open-Label Study of DCC-2618 to Assess Efficacy, Safety, and Pharmacokinetics In Patients With Advanced Gastrointestinal Stromal Tumors Who Have Progressed On Prior Anticancer Therapies.
Brief Title: A Study of DCC-2618 (Ripretinib) In Patients With With Advanced Gastrointestinal Stromal Tumors (GIST)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZL-2307-002
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-12

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumors,GIST,DCC-2618,Ripretinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — ripretinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- DCC-2618 (Experimental): DCC-2618 drug is 50mg per tablet, 150mg once a day, with 28 days as a treatment cycle.
  Interventions: Drug: DCC-2618

INTERVENTIONS:
Drug: DCC-2618 — Oral kinase inhibitor
  Other Names: Ripretinib

SUMMARY:
The primary objective of this trial is to evaluate the progress free survival (PFS) of DCC-2618 in patients with advanced gastrointestinal stromal tumors who have progressed with prior anticancer therapies based on independent radiologic review.

DETAILED DESCRIPTION:
The primary objective of this trial is to evaluate the progress free survival (PFS) of DCC-2618 in patients with advanced gastrointestinal stromal tumors who have progressed with prior anticancer therapies based on independent radiologic review. This study enrolled 39 subjects of 9 sites in China mainland, and all enrolled subjects received DCC-2618 after enrollment as treatment.

The study used EDC to collect patient data and IRT system for patient randomization, using Imaging Endpoints as the central image to evaluate the PFS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years of age.
* Patients with advanced gastrointestinal stromal tumors.
* Subjects who have progressed or documented intolerance after previous treatments.
* Sign informed consent, understand the Protocol and could follow the Protocol.
* The subject had at least one measurable lesion.
* Adequate organ function and bone marrow reserve

Exclusion Criteria:

* Treatment with anticancer therapy, including investigational therapy, or investigational procedures within 14 days or 5 x the half-life (whichever is longer) prior to the first dose of investigational drug.
* Prior treatment with DCC-2618.
* Previously or currently has an additional malignancy that is progressing or required active treatment, which may interfere with the safety or efficacy evaluation of DCC-2618.
* Patient has known active central nervous system metastases.
* New York Heart Association class II - IV heart disease, active ischemia or any other uncontrolled cardiac condition.
* Arterial thrombotic or embolic events within 6 months before the first dose of investigational drug.
* Venous thrombotic events within 3 months before the first dose of investigational drug.
* 12-lead electrocardiogram (ECG) demonstrating QT interval corrected by Fridericia's formula >450 ms in males or >470 ms in females at screening or history of long QT interval syndrome.
* Left ventricular ejection fraction (LVEF) <50% at screening.
* Use of known substrates or inhibitors of breast cancer resistance protein (BCRP) transporters within 14 days or 5 x the half-life (whichever is longer) prior to the first dose of investigational drug.
* Major surgeries within 4 weeks of the first dose of investigational drug.
* Any other clinically significant comorbidities, which in the judgment of the investigator, could compromise compliance with the protocol, interfere with interpretation of the study results, or predispose the patient to safety risks.
* Active viral infections.
* If female, the patient is pregnant or lactating, or plans to become pregnant during the study treatment period.
* Known allergy or hypersensitivity to any component of the investigational drug.
* Gastrointestinal abnormalities.
* Any active hemorrhages, excluding hemorrhoids or gum bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2022-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zai Lab, Study Director — Zai Lab (Shanghai) Co., Limited
Locations (9):
- China (9):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Union Medical College Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality
  - Union Medical College Hospital, Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2020 and August 2020, 39 patients were enrolled, and all received at least one dose of study drug.
Pre-assignment Details: 50 patients were assessed for eligibility, 11 experienced screen failure.
Period: Overall Study
Arm/Group | DCC-2618
Started | 39
Completed | 20 (20 participants died as of 30Aug 2022.)
Not Completed | 19
Not completed — Remained on treatment | 6
Not completed — Survival follow-up | 11
Not completed — Withdrawal of informed consent | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | DCC-2618
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 55.1 [36.8 to 73.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 39
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 39
ECOG performance status [Count of Participants; unit: Participants] — Patients with lower ECOG scores tend to have a relatively better prognosis.
  Participants
    0 | 7
    1 | 28
    2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS) is defined as the time from the first dose of study drug to the first occurrence of disease progression based on independent radiology review or death due to any cause (whichever occurred first).
Time Frame: Approximately 10 months since the first subject enrolled.
Population: Efficacy analyses were performed using the efficacy analysis set (EAS), consisting of the 38 participants who had received continuous ripretinib treatment since C1D1. 1 subject discontinued treatment due to clinical progression during the intensive blood sampling period and a total of 38 subjects who entered treatment period (continuous dose period) were included in the Efficacy Analysis Set (EAS).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | DCC-2618
Number analyzed (Participants) | 38
months | 6.44 [2.89 to 8.31]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The objective response rate (ORR) is defined as the percentage of participants who achieved confirmed complete response (CR) or partial responses (PR) based on independent radiology review.
Time Frame: Approximately 15 months since the first subject enrolled.
Population: 1 subject discontinued treatment due to clinical progression during the intensive blood sampling period and a total of 38 subjects who entered treatment period (continuous dose period) were included in the Efficacy Analysis Set (EAS).
Measure: Count of Participants; unit: Participants
Arm/Group | DCC-2618
Number analyzed (Participants) | 38
Participants | 8

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from the first dose of study drug to all-cause death.
Time Frame: Approximately 28 months since the first subject enrolled.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DCC-2618
Number analyzed (Participants) | 38
months | 25.56 [11.73 to NA] — The upper limit of 95% confidence interval was not estimated due to insufficient number of participants with events.

4. Secondary Outcome: Time to Best Response (TBR)
Description: Time to Best Response(TBR) based on independent radiology review is defined as the duration from the date of the first dose of the investigational drug to the date of confirming the best response.
Time Frame: Approximately 15 months since the first subject enrolled.
Measure: Median (Full Range); unit: months
Arm/Group | DCC-2618
Number analyzed (Participants) | 8
months | 2.25 [1.0 to 11.9]

5. Secondary Outcome: Disease Control Rate (DCR) (Confirmed CR + Confirmed PR + SD) for 12 Weeks
Description: Disease control rate (DCR) based on independent radiology review (confirmed CR + confirmed PR + SD for 12 weeks)
Time Frame: Approximately 15 months since the first subject enrolled.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DCC-2618
Number analyzed (Participants) | 38
Participants | 20

ADVERSE EVENTS:
Time Frame: From the date of the first dose of study treatment up to 30 days following study treatment discontinuation. Up to approximately 28 months.
Arm/Group | DCC-2618
All-Cause Mortality (participants affected / at risk) | 20/39
Serious Adverse Events (participants affected / at risk) | 10/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DCC-2618 (N=39)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 2
Pyrexia (General disorders) | 1
Cardiac dysfunction (Cardiac disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Acute myocardiac infarction (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
Inra-abdomina fluid collection (Gastrointestinal disorders) | 1
Aabdominal pain (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Interstitial lung desease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DCC-2618 (N=39)
Anaemia (Blood and lymphatic system disorders) | 26
Alopecia (Skin and subcutaneous tissue disorders) | 17
Asthenia (General disorders) | 13
Bilirubin conjugated increased (Investigations) | 13
Blood bilirubin increased (Investigations) | 13
Weight decreased (Investigations) | 10
Abdominal distension (Gastrointestinal disorders) | 9
Hypokalaemia (Metabolism and nutrition disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 7
Blood bilirubin unconjugated increased (Investigations) | 7
Blood creatine phosphokinase increased (Investigations) | 7
Sinus bradycardia (Cardiac disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Gamma-glutamyltransferase increased (Investigations) | 6
Lipase increased (Investigations) | 6
White blood cell count decreased (Investigations) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Aspartate aminotransferase increased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 5
Blood creatinine increased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 5
Headache (Nervous system disorders) | 5
Proteinuria (Renal and urinary disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Contrast media allergy (Immune system disorders) | 4
Urinary tract infection (Infections and infestations) | 4
Neutrophil count decreased (Investigations) | 4
Urinary occult blood positive (Investigations) | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Insomnia (Psychiatric disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4
Arrhythmia (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 3
Supraventricular extrasystoles (Cardiac disorders) | 2
Hypothyroidism (Endocrine disorders) | 3
Xerophthalmia (Eye disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Gingival bleeding (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Chest discomfort (General disorders) | 3
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 3
Hepatic pain (Hepatobiliary disorders) | 2
Folliculitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 3
Apolipoprotein A-I increased (Investigations) | 2
Apolipoprotein B increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 3
Blood creatine phosphokinase MB increased (Investigations) | 3
Blood fibrinogen increased (Investigations) | 3
Blood glucose increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 3
Blood urea increased (Investigations) | 2
C-reactive protein increased (Investigations) | 2
Coagulation test abnormal (Investigations) | 2
Glomerular filtration rate decreased (Investigations) | 2
High density lipoprotein increased (Investigations) | 2
Low density lipoprotein increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 2
Neutrophil count increased (Investigations) | 2
Protein urine present (Investigations) | 3
Red blood cells urine positive (Investigations) | 3
White blood cell count increased (Investigations) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT04282980/Prot_SAP_000.pdf